CLINICAL TRIAL: NCT01351064
Title: Using Computers to Assist in the Diagnosis and Treatment of Attention-deficit/Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Library of Medicine (NLM) (NIH)
Responsible Party: Principal Investigator, Aaron Carroll, Assoc. Prof of Pediatrics, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: CHICA_ADHD_Study; R01LM010031 (NIH)
Record Dates: First submitted 2011-05-09; First posted 2011-05-10 (Estimated); Results first posted 2015-12-18 (Estimated); Last update posted 2016-01-25 (Estimated); Status verified 2015-12

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CHICA ADHD Module (Experimental): This arm received The CHICA ADHD Module
  Interventions: Other: CHICA ADHD Module
- CHICA ADHD Control (No Intervention): This arm received CHICA without the ADHD module

INTERVENTIONS:
Other: CHICA ADHD Module — This module was added to CHICA to help diagnose and manage ADHD
  Arms: CHICA ADHD Module

SUMMARY:
Attention-deficit/hyperactivity disorder (ADHD) is the most commonly diagnosed behavioral disorder in children. Prevalence rates in the United States range from 2% to 18% depending on diagnostic criteria and population studied. Primary care physicians, especially pediatricians, have historically played a large role in the diagnosis and treatment of ADHD. Despite the existence of authoritative guidelines to assist primary care physicians, ample evidence demonstrates that they continue to diagnose and treat this disorder suboptimally. This is due, in part, to a lack of training and cumbersome delivery system designs. Modern computer decision support strategies offer the best hope of equipping general practitioners to deal with the mental health epidemic of ADHD.

The investigators have developed a novel decision support system for implementing clinical guidelines in pediatric practice. CHICA (Child Health Improvement through Computer Automation) combines three elements: (1) pediatric guidelines encoded in Arden Syntax; (2) a dynamic, scannable paper user interface; and (3) an HL7-compliant interface to existing electronic medical record systems. The result is a system that both delivers "just-in-time" patient-relevant guidelines to physicians during the clinical encounter, and accurately captures structured data from all who interact with it. Preliminary work with CHICA has demonstrated the feasibility of using the system to implement and evaluate clinical guidelines. The investigators propose to expand CHICA to include ADHD diagnosis and treatment guidelines. The investigators hypothesize that implementation of the ADHD guidelines will result in better outcomes, including higher rates of adherence to recommendations and improved patient functioning.

DETAILED DESCRIPTION:
Attention-deficit/hyperactivity disorder (ADHD) is the most commonly diagnosed behavioral disorder in children. Prevalence rates in the United States range from 2% to 18% depending on diagnostic criteria and population studied. Primary care physicians, especially pediatricians, have historically played a large role in the diagnosis and treatment of ADHD. Despite the existence of authoritative guidelines to assist primary care physicians, ample evidence demonstrates that they continue to diagnose and treat this disorder suboptimally. This is due, in part, to a lack of training and cumbersome delivery system designs. Modern computer decision support strategies offer the best hope of equipping general practitioners to deal with the mental health epidemic of ADHD.

The investigators have developed a novel decision support system for implementing clinical guidelines in pediatric practice. CHICA (Child Health Improvement through Computer Automation) combines three elements: (1) pediatric guidelines encoded in Arden Syntax; (2) a dynamic, scannable paper user interface; and (3) an HL7-compliant interface to existing electronic medical record systems. The result is a system that both delivers "just-in-time" patient-relevant guidelines to physicians during the clinical encounter, and accurately captures structured data from all who interact with it. Preliminary work with CHICA has demonstrated the feasibility of using the system to implement and evaluate clinical guidelines. The investigators propose to expand CHICA to include ADHD diagnosis and treatment guidelines. The investigators hypothesize that implementation of the ADHD guidelines will result in better outcomes, including higher rates of adherence to recommendations and improved patient functioning.

The specific research aims of this proposal are:

Aim 1: Expand and modify an existing computer-based decision support system (CHICA) to include ADHD treatment and diagnosis guideline rules as well as the capability to fax data directly into the medical record.

Aim 2: Evaluate the effect of the CHICA system on the processes of ADHD care in pediatric practices, including adherence to guidelines for ADHD treatment and diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Child between age 5 and 12 years seen in one of our clinics

Exclusion Criteria:

* Child outside the age range or who is not seen in one of our clinics.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 84 (Actual)
Dates: Start 2010-07; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron E Carroll, MD, MS, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Children's Health Services Research, Indianapolis, Indiana, United States

REFERENCES:
- [Derived] Carroll AE, Bauer NS, Dugan TM, Anand V, Saha C, Downs SM. Use of a computerized decision aid for ADHD diagnosis: a randomized controlled trial. Pediatrics. 2013 Sep;132(3):e623-9. doi: 10.1542/peds.2013-0933. Epub 2013 Aug 19. PMID 23958768

RESULTS

PARTICIPANT FLOW:
Groups:
- CHICA ADHD Module: This arm received The Child Health Improvement through Computer Automation (CHICA) Attention Deficit Hyperactivity Disorder (ADHD) Module
  CHICA ADHD Module: This module was added to CHICA to help diagnose and manage ADHD
Period: Overall Study
Arm/Group | CHICA ADHD Module | CHICA ADHD Control
Started | 42 | 42
Completed | 42 | 42
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CHICA ADHD Module | CHICA ADHD Control | Total
Number analyzed (Participants) | 42 | 42 | 84
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 42 | 42 | 84
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 11 | 24
  Male | 29 | 31 | 60
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 19 | 29 | 48
  White | 21 | 9 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Children Diagnosed With ADHD With Structured Diagnostic Assessment
Time Frame: one year
Measure: Number; unit: number of kids
Arm/Group | CHICA ADHD Module | CHICA ADHD Control
Number analyzed (Participants) | 42 | 42
number of kids | 34 | 16

2. Secondary Outcome: Percent of Patients Receiving ADHD Care Component
Time Frame: one year
Measure: Number; unit: percentage of participants
Arm/Group | CHICA ADHD Module | CHICA ADHD Control
Number analyzed (Participants) | 42 | 42
percentage of participants
  Medication adjusted | 45 | 33
  Reassessment of symptoms | 50 | 33
  Mental Health Referral | 74 | 55
  Mental Health Visit | 67 | 48

ADVERSE EVENTS:
Time Frame: Three months
Arm/Group | CHICA ADHD Module | CHICA ADHD Control
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/42
Other Adverse Events (participants affected / at risk) | 0/42 | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No